CLINICAL TRIAL: NCT03570671
Title: Dual-acquisition of Noninvasive Cardiac Imaging in Vasospastic Angina Korean Registry
Brief Title: Noninvasive Cardiac Imaging in Vasospastic Angina Korean Registry (NAVIGATOR)
Acronym: NAVIGATOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, Professor, Dept. of Cardiology, Dong-A University Hospital, Dong-A University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NAVIGATOR
Record Dates: First submitted 2018-05-29; First posted 2018-06-27 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Spasm
Keywords: MDCTA; Coronary artery spasm
MeSH Terms: conditions — Spasm; Coronary Vasospasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Spasm positive (Experimental): Ergonovine-induced coronary spasm provocation test positive: defined as transient, total, or sub-total occlusion (>90% stenosis) of a coronary artery with symptoms of myocardial ischemia (angina pain and ischemic ECG change).
  Interventions: Diagnostic Test: Spasm positive
- Spasm negative (Placebo Comparator): Suspected vasospastic angina subjects with negative ergonovine provocation test are considered as reference modality.
  Interventions: Diagnostic Test: Spasm negative

INTERVENTIONS:
Diagnostic Test: Spasm positive — Investigators define the positive criteria for VSA on MDCTA as follows:
  1. Significant stenosis (≥ 50%) with negative remodeling but no definite evidence of plaques, which completely dilated on IV nitrate CT, or
  2. Diffuse small diameter (< 2mm) of a major coronary artery with beaded appearance which completely dilated on IV nitrate CT.
  Arms: Spasm positive
Diagnostic Test: Spasm negative — Suspected vasospastic angina subjects with negative MDCTA-derived VSA are considered as reference modality.
  Arms: Spasm negative

SUMMARY:
With regard to the characteristics of spasm segment, had been clearly described by other invasive imaging methods including intravascular ultrasound and optical coherence tomography. However, there is potential risk during these invasive procedures, such as severe myocardial ischemia or fatal arrhythmia.

Presently available imaging test for coronary artery disease in multi detector-row computed tomography angiography (MDCTA) evaluation has high diagnostic accuracy to evaluate coronary artery stenosis. However, previous report assessing imaging findings or diagnostic accuracy of MDCTA in patients with vasospastic angina (VSA) is lacking.

DETAILED DESCRIPTION:
Previously investigators analyzed the characteristics of coronary spasm segment in an observational individual dataset, suspected VSA patients (n=20) underwent dual-acquisition of MDCTA (initial and intravenous nitrate injected CT imaging), the diagnostic accuracy showed sensitivity: 73%, specificity: 100%, positive predictive value: 100%, and negative predictive value: 56%.

Further study is necessary because previous analysis presented limited sample size and deficiency of healthy control.

Therefore, investigators hypothesis that dual-acquisition of MDCTA in noninvasive tool for coronary assessment provide more information of coronary characteristics, and the diagnostic efficacy would be non-inferior as compared with the invasive coronary imaging modality in coronary spasm-induced angina attacks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is onset of angina-like attack at rest, during effort, or during rest and effort.
* Subject has chest pain between night and early morning.
* Subject is scheduled to undergo MDCTA.
* Subject is an acceptable candidate for CAG with an EG provocation test.
* Cardiac condition: BP>90/60mmHg, ECG: sinus rhythm with regular, left ventricular ejection fraction>55%, and resting heart rate<100 beats/min.
* Subject will be provided written informed consent.
* Subject is willing to comply with study follow-up requirement.

Exclusion Criteria:

* Subject has clinical evidence of acute coronary syndrome.
* Subject has evidence of significant narrowing (>50% stenosis by CAG).
* Subject has clinical evidence of cardiomyopathy or valvular heart disease.
* Subject is hemodynamically unstable.
* Subject has a history of PCI and CABG.
* Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
* Subject has known allergy to contrast medium.
* Subject has renal insufficiency (serum creatine >2.5 mg/dl).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 3 days
  MDCTA procedure: all subjects will undergo MDCTA without a vasodilator ("initial CT") in the early morning before the ergonovine provocation spasm test. Subsequent "IV nitrate CT" will be allowed at a 3-day washout period after the first contrast usage. The scan protocol for the IV nitrate CT is as follows: during continuous injection of the intravenous vasodilating agent (isosorbidedinitrate 2 mg/hr), blood pressure will be checked every 2 minutes. When both the systolic and diastolic blood pressure decrease by 10 mmHg in comparison to the initial value, the CT scan initiate and images will be acquired during the nitrate infusion.
  Investigators define the positive criteria for VSA on MDCTA as follows:
  1. Significant stenosis (≥ 50%) with negative remodeling but no definite evidence of plaques, which completely dilated on IV nitrate CT, or
  2. Diffuse small diameter (< 2mm) of a major coronary artery with beaded appearance which completely dilated on IV nitrate CT.

SECONDARY OUTCOMES:
Coronary vessel distensibility | 3 days
  To evaluate the extent of coronary vessel distensibility by dual-acquisition of cardiac MDCTA in patients with VSA
Cutoff value of coronary vessel distensibility index | 3 days
  To consider the cutoff value of coronary vessel distensibility index (CVDI) to predict the coronary spasm induced angina-like attacks.
  Investigators define the CVDI as following formulas:
  1. CVDI-CSA (cross-section area)= [(CSA_IV nitrate - CSA_initial) / CSA_IV nitrate]ⅹ100% or
  2. CVDI-D (diameter)= [(D_IV nitrate - D_initial) / D_IV nitrate]ⅹ100%.
Incidence of multi-vessel spasm | 3 days
  To examine the incidence of multi-vessel coronary spasm by MDCTA.
Diagnostic accuracy of MDCTA | 3 days
  To determine the diagnostic accuracy of MDCTA modalities for detection of VSA.
Characteristics of spasm-related coronary artery segment | 3 days
  To describe the characteristics of spasm-related coronary artery segment including vessel remodeling, plaque composition and stenosis degree.

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, MD, Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang EJ, Kim MH, De Jin C, Seo J, Kim DW, Yoon SK, Park TH, Lee KN, Choi SI, Yoon YE. Noninvasive detection of coronary vasospastic angina using a double-acquisition coronary CT angiography protocol in the presence and absence of an intravenous nitrate: a pilot study. Eur Radiol. 2017 Mar;27(3):1136-1147. doi: 10.1007/s00330-016-4476-2. Epub 2016 Jul 6. PMID 27380904
- [Background] Jin C, Kim MH, Kang EJ, Cho YR, Park TH, Lee KN, Serebruany V. Assessing Vessel Tone during Coronary Artery Spasm by Dual-Acquisition Multidetector Computed Tomography Angiography. Cardiology. 2018;139(1):25-32. doi: 10.1159/000478926. Epub 2017 Nov 23. PMID 29166637